CLINICAL TRIAL: NCT00388050
Title: Wiser Choices for Patients With Type II Diabetes: Diabetes Medication Choice
Brief Title: Diabetes Medication Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Victor Montori, Mayo Clini
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-003513; ADA #33
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
Keywords: Decision aid, diabetes, primary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Diabetes Medication Choice decision aid (Experimental): Patients in this arm will discuss diabetes medication for glucose control with the help of a decision aid that covers five commonly prescribed anti-hyperglycemic medications.
  Interventions: Behavioral: Diabetes Medication Choice decision aid
- Usual Care (Other): Patients and clinicians in this arm will discuss anti-hyperglycemic agents in their usual manner.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Diabetes Medication Choice decision aid — The decision aid covers five commonly prescribed anti-hyperglycemic medications and their attributes.
  Arms: Diabetes Medication Choice decision aid
Behavioral: Usual Care — Patients and clinicians in this arm will discuss anti-hyperglycemic agents in their usual manner.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to examine how different ways of sharing information about diabetes medication treatment options with patients can affect their choices and health.

ELIGIBILITY:
* Have a diagnosis of type 2 diabetes mellitus of any duration; c-peptide test not required
* Use 1 or 2 oral hypoglycemic agents; not using insulin therapy
* Are not pregnant
* Have stable but inadequate glycemic control: both A1C at the time of eligibility and previous A1c within 6 months between 7-9.5%
* Recognize their primary care provider as their main diabetes care provider
* Do not have major barriers (i.e., severe hearing impairment, dementia, cannot communicate in English) to participate in shared decision-making (per provider?s assessment)
* Have no plans to relocate out of town in the next 6 months
* Enrolment is open to males and females of diverse racial backgrounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Understanding | Directly proceeding the clinical encounter
Decisional Conflict | Directly proceeding the clinical visit
Treatment Action, adherence | Directly proceeding the clinical encounter, 6 months after the clinical encounter

SECONDARY OUTCOMES:
Trust | Directly proceeding the clinical visit
Acceptability | Directly proceeding the clinical encounter

CONTACTS AND LOCATIONS:
Overall Officials: Victor M. Montori, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289
- [Derived] LeBlanc A, Ruud KL, Branda ME, Tiedje K, Boehmer KR, Pencille LJ, Van Houten H, Matthews M, Shah ND, May CR, Yawn BP, Montori VM. The impact of decision aids to enhance shared decision making for diabetes (the DAD study): protocol of a cluster randomized trial. BMC Health Serv Res. 2012 May 28;12:130. doi: 10.1186/1472-6963-12-130. PMID 22640439
- [Derived] Mullan RJ, Montori VM, Shah ND, Christianson TJ, Bryant SC, Guyatt GH, Perestelo-Perez LI, Stroebel RJ, Yawn BP, Yapuncich V, Breslin MA, Pencille L, Smith SA. The diabetes mellitus medication choice decision aid: a randomized trial. Arch Intern Med. 2009 Sep 28;169(17):1560-8. doi: 10.1001/archinternmed.2009.293. PMID 19786674